CLINICAL TRIAL: NCT03215108
Title: Comparison Between Novel Flower-type Covered Stent and Conventional Covered Stent in Malignant Extrahepatic Biliary Obstruction: Prospective Randomized Multicenter Study
Brief Title: Comparison Between Novel Flower-type Covered Stent and Conventional Covered Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-03-098-001
Record Dates: First submitted 2017-05-26; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-05

CONDITIONS: Malignant Biliary Obstruction
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Intervention Model Description: Flower-CSEMS vs. Conventional-CSEMS
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flower-CSEMS (Experimental): EGIS Flower Biliary Full Covered Stent(Flower-CSEMS), Bile Duct Stent, (S & G Biotech Co., Ltd.) will be inserted by using Endoscopic Retrograde CholangioPancreatography(ERCP).
  Interventions: Device: Endoscopic Retrograde CholangioPancreatography(ERCP)
- Conventional-CSEMS (Experimental): Conventional-CSEMS (S & G Biotech Co., Ltd.) will be inserted by using Endoscopic Retrograde CholangioPancreatography(ERCP).
  Interventions: Device: Endoscopic Retrograde CholangioPancreatography(ERCP)

INTERVENTIONS:
Device: Endoscopic Retrograde CholangioPancreatography(ERCP) — This study is prospective randomized multicenter study by using Endoscopic Retrograde CholangioPancreatography(ERCP). Comparison between Novel flower-type covered stent and Conventional covered stent in malignant extrahepatic biliary obstruction will be conducted after stent insertion by using Endoscopic Retrograde CholangioPancreatography(ERCP).

SUMMARY:
The aim of this animal study is determining the technical feasibility of the novel flower-type covered self-expandable metal stent (F-CSEMS) and investigating whether the novel flower-type covered self-expandable metal stent (F-CSEMS) could prevent cholecystitis and pancreatitis, comparing with conventional covered self-expandable metal stent (C-CSEMS).

DETAILED DESCRIPTION:
Covered self-expandable metal stent (C-CSEMS) has the risk of obstruction of the cystic duct, and the main and branch pancreatic ducts due to strong radial force and covering material, which results in cholecystitis and pancreatitis.

A flower-type covered self-expandable metal stent (F-CSEMS) having a five-petal-shaped design with side grooves was constructed to prevent the obstruction of the cystic duct orifice.

This study investigated the value of the F-CSEMS in protection for cholecystitis and pancreatitis.

The investigators will enroll patients with distal MBO (Malignant Biliary Obstruction) who received placement at the Samsung Medical Center. Transpapillary flower-type covered self-expandable metal stent (F-CSEMS) placements will be included in this study.

The diagnosis of MBO will be based on imaging and/or pathological findings. Malignancy was proved by histopathological confirmation obtained by endoscopic ultrasonography-guided fine-needle aspiration (EUS-FNA), bile duct biopsy (cytology), pancreatic duct cytology, or liver biopsy.

The investigators will evaluate the frequency of pancreatitis and cholecystitis.

Furthermore, the investigators will evaluate various parameters to clarify the predictive factors of pancreatitis and cholecystitis. The following 10 variables will be evaluated in pancreatitis by univariate analysis: [1] sex, [2] age, [3] primary disease, [4] Covered type (partially or fully), [5] SEMS with high AF, [6] F-CSEMS with high RF, [7] EST before F-CSEMS, [8] previous biliary stent, [9] contrast injection into the pancreatic duct (pancreatogram), and [10] the position of the distal stent edge.

The following 11 variables will be evaluated in cholecystitis by univariate analysis: [1] sex, [2] age, [3] regions of stricture, [4] F-CSEMS with high AF AF (axial force), [5] F-CSEMS with high RF, [6] previous biliary stent, [7] gallbladder stone, [8] contrast injection into the gallbladder (GB injection), [9] involvement to the orifice of the cystic duct (OCD), [10] position of distal stent edge, and [11] cystic duct occlusion by F-CSEMS.

--------------------------------------------------------------------------------------------------------

software: nQuery + nTerim (version 4.0)

- One-sided Chi-square test for proportion comparison

H0: p1=p2 vs H1: p1>p2 (The incidence of complications in the flower-type covered stent is smaller than in the conventional stent.)

p1 = incident rate of complication in full covered stent group p2 = incident rate of complication in flower-type covered stent group

* Set p1(incident rate of complication in full covered stent group) = 15% = 0.15
* expected % decrement in incidence rate = 40%, 50%, 60%, 70% --> p2 = 0.09, 0.075, 0.06, 0.045
* Significance level (alpha) = 0.05
* Maximum number of patients who can be enrolled = 10 per month at SMC = 120 per year
* Expected enroll period = 1 year = 12 months

  1. Sample size calculation with targeted power of 80% Expected % decrement in incidence rate 70% p2 4.5% Required n per group 116 Required total sample size 232 Required enroll period (year) 1.9
  2. Power calculation with a total sample size of 232 (116 per group) Expected % decrement in incidence rate 40% 50% 60% 70% p2 9.0% 7.5% 6.0% 4.5% Expected power (%) 32 48 64 80
  3. Minimum % decrement to be detected with power of 80% Planned enroll period (year) 1 1.5 2 2.5 3 Enroll-able n per group 60 90 120 150 180 Enroll-able total sample size 120 180 240 300 360 Minimum % decrement to be detected 93.33% 78.70% 68.70% 62.70% 58.00% Expected p2 1.0% 3.2% 4.7% 5.6% 6.3%

ELIGIBILITY:
Inclusion Criteria:

* Adults from 19 to 85 years of age who have voluntarily agreed to the clinical trial and signed a written agreement
* Patients with malignant extrahepatic bile duct obstruction without surgery

Exclusion Criteria:

* Patients who had already undergone surgical biliary drainage
* Patients who previously underwent percutaneous spinal cholecystectomy (PTGBD)
* Patients who underwent conventional metal-on-metal self-expandable metal stents (C-CSEMS)
* Patients who underwent biliary plastic stent implantation for more than 15 days
* Patients with malignant stricture of the intrahepatic bile duct and patients with stenosis within 2 cm of the liver
* Patients whose expected life expectancy is less than 3 months
* Pregnant patient
* Patients who can not undergo endoscopic procedures based on the judgment of the researcher

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2017-07-12 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pancreatitis, Cholecystitis - Occurrence rate : % | 3 months after procedure
  The incidence of pancreatitis is calculated using percentiles.
Pancreatitis, Cholecystitis - Severity | 3 months after procedure
  The extent of each side effect is described in the Adverse Reactions Report according to the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) Rating System version 4.0.

SECONDARY OUTCOMES:
Stent-related adverse events | 6 months after procedure
  Post -ERCP pancreatitis, Severity of pancreatitis, Bleeding, Microperforation
Stent patency | 6 months after procedure
  We followed up the stent patency until the time of patient death or stent occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Kyun Lee, MD PhD, Study Chair — Samsung Medical Center
Locations (1):
- SamsungMC, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No